CLINICAL TRIAL: NCT05895734
Title: Effectiveness of Upper Limb Rehabilitation Using the Powerball System in People With Multiple Sclerosis
Brief Title: Effectiveness of Powerball System in People With Multiple Sclerosis
Acronym: EMPOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EM_POWERBALL23
Record Dates: First submitted 2023-05-25; First posted 2023-06-09 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Neurologic Disorder; Multiple Sclerosis
MeSH Terms: conditions — Nervous System Diseases; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powerball (Experimental): Rehabilitation using the Powerball system
  Interventions: Device: NDS-Powerball®,
- Conventional treatment (Active Comparator): Rehabilitation by conventional treatment
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: NDS-Powerball®, — Rehabilitation using the Powerball system
  Arms: Powerball
Other: Conventional treatment — Rehabilitation by conventional treatment
  Arms: Conventional treatment

SUMMARY:
There is a high percentage of impairment in the upper limbs (UL) in patients with multiple sclerosis (MS), being muscle strength and hand dexterity a determining factor for the preservation of functional activities, constituting the basis of independence and quality of life. The aim of this study is to determine the effects of a training protocol on UL muscle strength, through the NDS-Powerball® system, in combination with conventional physiotherapy, during 8 weeks in terms of muscle strength, coordination, fatigue, functionality and quality of life in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years
* Diagnosed with MS according to McDonald criteria with an evolution time of more than two years
* Evaluation in the Kurtzke Disability Status Scale in Multiple Sclerosis (EDSS) with a score between 3.5 and 6
* Score less than or equal to 4 on the "Pyramidal Function" section of the EDSS functional scale
* Stable medical treatment for at least six months prior to surgery
* Muscle tone in the upper extremities no greater than 2 points on the modified Ashworth scale.
* Muscle balance equal to or greater than 3 in the upper extremity
* Absence of cognitive impairment with ability to understand instructions and score equal to or greater than 4 on the Minimental Test.

Exclusion Criteria:

* Diagnosis of another neurological disease or musculoskeletal alteration other than MS
* Diagnosis of any cardiovascular, respiratory or metabolic disease or other conditions that may interfere with this study
* Having suffered an exacerbation or hospitalization in the last three months before starting the assessment protocol, or during the therapeutic intervention process.
* Having received treatment with botulinum toxin in the six months prior to the start of the study
* Presence of visual alterations not corrected by means of ocular devices.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Isometric hand strength: | 1 minute
  Measured through the JAMAR® fist dynamometer, which is a sealed hydraulic system with an adjustable space to adapt to the handgrip of each patient. The JAMAR® dynamometer has been widely cited and is considered the gold standard for the assessment of handgrip strength. In turn, its test-retest and inter-rater reliability is excellent in different populations. The patient held the tool with the upper limb at 0º of abduction and rotation; elbow flexed at 90º and the forearm in neutral position; wrist between 0 and 15º of radial deviation; and performed a maximum grip for 3 seconds with his 5 fingers, quantifying the force exerted in kilograms. Three measurements were taken with each hand, always starting with the dominant hand; once the three measurements were taken, the mean of these was used.
Isometric pincer force | 3 minutes
  A Baseline Pinch Gauge® was used to assess pinch force. Three presses were performed with the maximum possible force for 3 seconds, alternating between the dominant and non-dominant hand; the force obtained is marked in kilograms by the dynamometer. Once the 3 results were obtained, the average of these was obtained.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | 3 minutes
  used to assess coordination and manual dexterity. The patient is seated with the tool, a wooden box divided into two identical halves inside which there are 150 cubes of 2.5 cm of wood of different colors, in front of his midline. The patient has to pass as many cubes as possible from one half of the box to the other in 60 seconds. The test is performed first with the dominant hand and then with the non-dominant hand. It is a standardized tool for the measurement of the gross function of the MMSS, having been validated by gender and age in healthy subjects, in turn, it shows a low ceiling and floor effect in people with MS. On the other hand, other psychometric properties such as test-retest reliability and minimum detectable change have been studied in other neurological pathologies, the former being excellent and the latter finding its cut-off point in 6 blocks.
Nine Hole Peg Test (NHPT) | 2 minutes
  this test was used to assess the function of the upper limbs, in particular fine motor skills of the hand. The tool is placed in front of the subject's midline, the subject has to insert the 9 pegs, one at a time, into the 9 holes of a board and then remove them, again one at a time, in the shortest possible time; first with the dominant hand, and then the non-dominant hand, the hand that is not being assessed can hold the board to provide stability. The score is the time in seconds required to insert and remove all the pins. It shows excellent test-retest, inter-rater and inter-rater reliability and adequate internal consistency. Scores above 0.27 seconds per pin indicate severe hand dysfunction. The minimum detectable change for the non-dominant hand is 7.46 seconds, while for the dominant hand it is 4.38 seconds. The standard error of measurement for the non-dominant hand is found to be 2.69 seconds, while for the dominant hand it is found to be 1.58 seconds
Abilhand test | 3 minutes
  is a self-completed questionnaire to assess the manual dexterity of the person, defining this as the ability to perform a series of tasks, regardless of the strategies applied to achieve it. It was originally developed for people with rheumatoid arthritis, and has subsequently been validated for different pathologies. The questionnaire contains 23 items, which correspond to various tasks of ADLs, the patient will mark the degree of difficulty he/she refers to when performing the activities, with 4 possible answers, "impossible", "difficult", "easy" and "not applicable", giving a score of 0, 1 and 2 points respectively, those activities that have not been performed in a period greater than or equal to 3 months will be not applicable. The score can range from 0 to 46 points, the higher the score, the better the manual dexterity. Its inter- and intra-rater reliability, internal consistency and construct validity are excellent.
Fatigue Severity Scale (FSS) | 2 minutes
  this is a self-applied scale that assesses the appearance of fatigue in the patient when performing certain daily activities. It has 9 items whose weighting ranges from 1 to 7, with 1 point being "completely disagree" and 7 points "completely agree". The minimum score is 9 points and the maximum score is 63. A higher score determines that fatigue interferes more with the patient's life. The standard error of measurement is 0.7 points. The minimum detectable change is 1.9 points. The test-retest reliability is moderate, and the construct validity is excellent for people with MS.
Multiple Sclerosis Impact Scale (MSIS-29) | 3 minutes
  is a self-applied scale on the impact of the disease on the patient's life in the two weeks prior to performing. It presents 29 questions of which 20 assess the physical aspects of MS and 9 assess the psychosocial aspects. There are 5 possible answers that score from 1 to 5 from least to most impact of the disease. Two total scores are generated corresponding to the physical and psychological impact subscales. The scoring range is from 0 to 100, with a higher score indicating a greater degree of disability. It was designed to be a scientifically rigorous, clinically useful and disease-specific instrument. The physical sphere has been proven to have high internal consistency and good construct validity, while the cognitive sphere has good internal consistency. Low ceiling and floor effects and an excellent Cobranch's Alpha for both parts of the scale and a strong correlation between both parts of the scale
Customer Satisfaction Questionnaire (CSQ8) | 2 minutes
  8-item questionnaire on the opinion of the attention or service perceived during the study. The score ranges from 1 to 4, these scores being "bad", "fair", "good" and "excellent". The higher the score, the greater the degree of satisfaction with the service
Likert satisfaction questionnaire for the experimental group | 1 minute
  at the end of the study, the participants in the experimental group also completed a satisfaction survey in relation to the experimental treatment carried out, using a Likert-type questionnaire prepared by the research team. This was a 20-item questionnaire on user satisfaction with the system used, ranging from attributes of the tool itself, ease of use or accessibility; design of the sessions, schedules, duration; as well as attributes of the center and physiotherapist involved in the intervention. The scores ranged from 1 to 5 points, with 1 point being "dissatisfied", 2 "not very satisfied", 3 "indifferent", 4 "satisfied", 5 "very satisfied".

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes